CLINICAL TRIAL: NCT05898360
Title: Promoting Immune Health by Intermittent
Brief Title: Promoting Immune Health by Intermittent Fasting: a Pilot Study
Acronym: TIGER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Max Nieuwdorp, professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2022.0697
Record Dates: First submitted 2023-02-12; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Metabolic Syndrome; HEALTHY VOLUNTEERS; Time Restricted Feeding; Insulin Resistance; Inflammation
MeSH Terms: conditions — Metabolic Syndrome; Intermittent Fasting; Insulin Resistance; Inflammation

STUDY DESIGN:
Intervention Model Description: daily time-restricted eating (TRE) protocol and a control protocol for each two weeks, separated by a four-week wash-out period
Who Masked: Outcomes Assessor
Masking Description: Investigators analysing study outcomes will be blinde
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- daily time-restricted eating (TRE) for 2 weeks (Experimental): Subjects will be instructed to consume all calories needed for a stable weight (based on their resting energy expenditure) in either one meal per day (TRE; between 10:00-11:00; a protein snack at 13 h) or in three meals per day (control; breakfast, lunch and dinner). Prior to the intervention, a dietician will instruct subjects on nutritional intake based on their caloric need measured by indirect calorimetry (see indirect calorimetry). During the intervention, subjects will fill in online or written dietary diary (e.g. eetmeter) and a physical activity diary. Halfway the intervention, a telephone consult with a dietician will take place
  Interventions: Combination Product: Time Restricted Eating
- control protocol for each two weeks (Placebo Comparator): Subjects will be instructed to consume normal diet/calories. Prior to the intervention, a dietician will instruct subjects on nutritional intake based on their caloric need measured by indirect calorimetry (see indirect calorimetry). During the intervention, subjects will fill in online or written dietary diary (e.g. eetmeter) and a physical activity diary. Halfway the intervention, a telephone consult with a dietician will take place
  Interventions: Other: normal diet

INTERVENTIONS:
Combination Product: Time Restricted Eating — time restricted eating
  Arms: daily time-restricted eating (TRE) for 2 weeks
Other: normal diet — normal diet
  Arms: control protocol for each two weeks

SUMMARY:
The goal is to study the direct effects of long-term intermittent fasting on immune cell populations in the blood, combined with analyses of systemic metabolic fitness and inflammatory activation of leukocytes.

DETAILED DESCRIPTION:
the investigators aim to investigate the direct effects of intermittent fasting on the molecular characteristics of monocytes and their related health benefits. In addition,the investigators want to assess the post-prandial inflammation and the potential protective role of IF on post-prandial monocyte activation and its related health benefits. This pilot study may better understand the molecular mechanisms behind IF, which could further personalize lifestyle guidance and identify novel anti-inflammatory processes that control immune responses and inflammation.

ELIGIBILITY:
Inclusion Criteria metsyn:

* BMI 30 to 43 kg/m2
* HOMA-IR index larger/same as 2.5
* And At least 3 out of 5 NCEP (National Cholesterol Education Program) metabolic syndrome criteria:
* Fasting plasma glucose ≥ 6.1 mmol/l,
* Triglycerides≥1.7mmol/l,
* Waist-circumference>102cm,
* HDL-cholesterol<1.04mmol/l,
* Bloodpressure≥130/85mmHg).

Inclusion healthy volunteers

* Body mass index (BMI) 18 to 25 kg/m2,
* Waist circumference between 79 cm and 94 cm and
* HOMA-IR index: ≤ 2.0 (measured as fasting insulin (pmol/L) x fasting glucose (mmol/L)) / 135)

Exclusion criteria; (all)

* Excessive weight loss of >10% in the last months;
* Use of any medication, including proton pomp inhibitors and antibiotics in the past three months;
* Cholecystectomy;
* Untreated GI disease/abnormal bowel habits;
* Plasma aspartate aminotransferase and alanine aminotransferase are 2.5 times or more the upper limit of the normal range;
* A history of cardiovascular event (MI or pacemaker implantation);
* A history of heavy alcohol use (>12 to 15 g of alcohol per day, or >12 oz of beer, 5 oz of wine, or 1.5 oz of distilled spirits);
* A dependency on alcohol or unable to pause the consumption of alcohol during the study period.
* An (expected) prolonged compromised immunity (due to recent cytotoxic chemotherapy or HIV infection with a CD4 count < 240);
* Unmotivated or not able to adhere to a specific diet;
* History of eating disorder;
* Night workers or people with deviant day/night rhythm;
* Pregnant, trying to get pregnant or breast feeding at inclusion;
* Irregular menstrual cycle;
* Hormonal replacement therapy (other than oral contraceptives).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-02-27 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Immune health | 0-2 weeks
  measured by transcriptomic assays for immune phenotyping
inflammatory activation of leukocytes | 0-2 weeks
  measured by flow cytometry

SECONDARY OUTCOMES:
Changes in post-prandial bile acid metabolism | 2 hours
  area under the curve of bile acid concentrations
The effect of IF on glucose tolerance | 2 hours and 0-2 weeks
  measured during high fat meal test as well during the inverention (by FSL)
The effect of IF on the transcriptional and epigenetic repertoire of whole blood monocytes by stimulation assays | 0-2 weeks
  the effect on the inflammatory status
The effect on energy expenditure | 2 hours
  resting energy expenditure measured by indirect calorimetry during high fat meal test
The effect of Impaired fasting on gut microbiota composition. | 0-2 weeks
  measured at the end of the intervention by 16S sequencing
Effect on Body composition and Appetite (visual analog scale scores + quantity of food consumed) | 0-2 weeks
  measured during high fat meal test in terms of fat mass(kg) and fat free mass (kg)
effect on appetie | 0-2 weeks
  visual scale scores (0(worst)-100%(best)) and quantity of food consumed

CONTACTS AND LOCATIONS:
Overall Officials: Maarten R Soeters, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No